CLINICAL TRIAL: NCT04316897
Title: Prevalence of Rheumatic Heart Disease According to Revised Jones Criteria (2015) in Assiut Governate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shady Hossam Nader Kamel, Principal investigator, Assiut University
Other Study IDs: LAPRHFP
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Rheumatic Fever
MeSH Terms: conditions — Rheumatic Fever | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Echocardiography — It is a an observational cross-sectional echocardiographic screening study in Assiut Governate conducted after seeking approval from the local institutional review board and human subjects' protection.

SUMMARY:
Prevalence of rheumatic heart disease according to revised jones criteria (2015) in Assiut governate

DETAILED DESCRIPTION:
Although acute rheumatic fever (ARF) has declined in Europe and North America in incidence over the past 4 to 6 decades, the disease remains one of the most important causes of cardiovascular morbidity and mortality especially in the developing countries that are home to the majority of the world's population(1), Incidence rates in these countries still reach epidemic levels(2).

In general, most patients with RHD do not have documented histories of ARF, and they present with late complications, such as heart failure, arrhythmia, stroke, endocarditis, or pregnancy-related complications(3).

Echocardiographic screening according to revised jones criteria (2015) (1) is the most reliable way of detecting RHD in asymptomatic people, and it can identify large numbers of previously undetected cases(4-6).

People with RHD detected by screening can receive appropriate cardiac care, including guideline-recommended secondary prophylaxis(7). This may be a cost-effective approach to managing RHD in groups at high risk in Assiut Governate(8). Nevertheless, large scale screening has not been undertaken, and studies are underway to determine the best models for sustainable targeted screening and to evaluate the impact of screening and treatment on clinical outcomes(9).

In this study, we aimed to determine the role of echocardiographic screening for detecting undiagnosed RHD, and to estimate the prevalence of RHD in Assiut Governate.

ELIGIBILITY:
Inclusion Criteria:

- Children and young adults aged 5-18 years living in Assiut Governate ,who are attending general clinics of Assiut University Children Hospital, were invited to participate in echocardiographic screening for RHD in February and October 2021. Informed consent will be obtained in writing from participants or their parents after providing explanations of the study in local languages.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study will be conducted in February and October 2021. It will include 384 children attending in outpatient general clinics of Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The aim of the study is to assess the prevalence of rheumatic heart disease (RHD) according to the American Heart Association modified Jones criteria 2015 (1). Cases will be defined as definite, probable or not RHD. | Baseline
  Prevalence of rheumatic heart disease according to revised jones criteria (2015) in Assiut governate Cases will be defined as definite, probable or not RHD. So, it will provide a great outcome for all the targeted patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fahim M. Fahim, Study Director — Doctor
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Gewitz MH, Baltimore RS, Tani LY, Sable CA, Shulman ST, Carapetis J, Remenyi B, Taubert KA, Bolger AF, Beerman L, Mayosi BM, Beaton A, Pandian NG, Kaplan EL; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young. Revision of the Jones Criteria for the diagnosis of acute rheumatic fever in the era of Doppler echocardiography: a scientific statement from the American Heart Association. Circulation. 2015 May 19;131(20):1806-18. doi: 10.1161/CIR.0000000000000205. Epub 2015 Apr 23. PMID 25908771